CLINICAL TRIAL: NCT06932874
Title: Study on the Efficacy and Safety of Metformin Hydrochloride Dicarboxylate Sustained-release Tablets (Ⅲ) in Patients With Type 2 Diabetes Mellitus Complicated With Coronary Heart Disease: An Open, Randomized Controlled Trial
Brief Title: Metformin Hydrochloride Sustained-release Tablets (Ⅲ) in Patients With Type 2 Diabetes Mellitus Complicated With Coronary Heart Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0408
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Heart Disease; Type 2 Diabetes
Keywords: Type 2 diabetes; coronary atherosclerotic heart disease; metformin hydrochloride sustained-release tablets (Ⅲ)
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucophage (Metformin Hydrochloride Tablets) (Active Comparator): Metformin hydrochloride tablets combined with other oral hypoglycemic drugs for 24 weeks treatment.
  Interventions: Drug: Glucophage (Metformin Hydrochloride Tablets)
- New type of metformin sustained-release tablets (Ⅲ) (Experimental): The experimental group received treatment with New Metformin Sustained-release Tablets (Ⅲ) combined with other oral hypoglycemic drugs for 24 weeks.
  Interventions: Drug: New sustained-release metformin tablets (Ⅲ)

INTERVENTIONS:
Drug: Glucophage (Metformin Hydrochloride Tablets) — Metformin hydrochloride tablets combined with other oral hypoglycemic drugs for 24 weeks treatment.
  Arms: Glucophage (Metformin Hydrochloride Tablets)
Drug: New sustained-release metformin tablets (Ⅲ) — The experimental group received treatment with New Metformin Sustained-release Tablets (Ⅲ) combined with other oral hypoglycemic drugs for 24 weeks.
  Arms: New type of metformin sustained-release tablets (Ⅲ)

SUMMARY:
The purpose of this study is1. Compare the differences in the changes of glycated hemoglobin after 24 weeks of treatment between the new metformin sustained-release tablets (Ⅲ) group and the metformin ordinary tablets group.

2. Compare the differences in the changes of fasting blood glucose, gastrointestinal adverse reactions of the drug and compliance after 24 weeks of treatment between the new metformin sustained-release tablets (Ⅲ) group and the metformin ordinary tablets group.

DETAILED DESCRIPTION:
A total of 356 patients with type 2 diabetes mellitus complicated with coronary heart disease were selected. According to the usage of oral hypoglycemic drugs before enrollment, they were divided into the group without using hypoglycemic drugs, the single-drug group (SGLT2i), and the dual-drug group (SGLT2i + DPP4i). Within the same group of subjects, they were randomly divided into the treatment group with the new metformin sustained-release tablets (Ⅲ) (referred to as the experimental group) and the control group with Glucophage (referred to as the control group) at a ratio of 1:1 for 24 weeks of intervention.

Outpatient follow-ups were conducted at baseline, 12 weeks, and 24 weeks, and the differences in glycated hemoglobin, fasting blood glucose changes, gastrointestinal adverse reactions, and compliance were compared between the two groups.

Telephone follow-ups were conducted at 4 weeks, 8 weeks, 16 weeks, and 20 weeks to compare the differences in fingertip blood glucose, gastrointestinal adverse reactions, and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 - 75 years old; BMI: 18.5 - 35 kg/m²
* T2DM meets the WHO standards of 1999, with HbA1c ranging from 7% to 9%, and fasting blood glucose ranging from 7 to 10 mmol/L.

  1. Newly diagnosed T2DM patients who only receive dietary control and exercise therapy
  2. T2DM patients who have been diagnosed before, with HbA1c still not reaching the standard after oral hypoglycemic drug treatment for at least 12 weeks, and the oral hypoglycemic drugs include two types: dipeptidyl peptidase-4 inhibitors (DPP-4i) and sodium-glucose cotransporter 2 inhibitors (SGLT2i), and have taken these drugs for at least 4 weeks.
* Before admission or during this admission, coronary heart disease was diagnosed by coronary angiography, and standard coronary heart disease routine treatment was carried out, including standard antiplatelet therapy, lipid-lowering therapy, and control of ventricular rate. Beta-blockers were uniformly treated with metoprolol sustained-release tablets, and antiplatelet drugs were uniformly treated with aspirin to avoid the influence of coronary heart disease drugs on hypoglycemic effects.

Exclusion Criteria:

* Within 4 weeks prior to enrollment, used glucagon-like peptide-1 receptor agonists (GLP-1RA) or metformin.
* Within 4 weeks prior to enrollment, had acute coronary syndrome, severe heart disease other than coronary artery disease, or chronic heart failure (NYHA IV grade).
* Patients who had failed PCI, planned staged revascularization, or had other types of stent implantation in the past.
* Patients with acute or chronic pancreatitis, severe neurological diseases, renal dialysis, advanced liver disease, other tumors, organ transplant post-operation, patients with a history of hormone therapy.
* Special types of diabetes, and endocrine diseases such as hyperthyroidism, hypothyroidism, primary aldosteronism, pheochromocytoma, Cushing's syndrome, congenital adrenal cortical hypofunction, pituitary tumor and hypopituitarism, multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma family or personal history, personal history of non-familial medullary thyroid carcinoma.
* Pregnant, in the process of pregnancy or lactation during the postpartum period.
* Within the past 12 weeks, had acute or chronic infectious diseases, fever, anemia, dehydration and electrolyte imbalance, elevated blood lactate level (reaching 2-4 mmol/L).
* Had lactate acidosis in the past (blood lactate ≥ 5 mmol/L, pH value ≤ 7.35 (arterial blood)).
* Liver and kidney dysfunction, with alanine aminotransferase and aspartate aminotransferase ≥ 3 times the upper limit, glomerular filtration rate ≤ 45 ml/min/min.
* Had esophageal reflux, gastric bleeding, peptic ulcer or other severe gastrointestinal diseases within the past 12 weeks.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline, 12 weeks, 24 weeks
  Glycated hemoglobin (HbA1c) at baseline, 12 weeks and 24 weeks through venous blood samples

SECONDARY OUTCOMES:
Fasting blood glucose | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks
  Baseline, 12 weeks, 24 weeks samples were collected by venous blood draw; while 4 weeks, 8 weeks, 16 weeks and 20 weeks samples were collected by fingertip blood draw.
Gastrointestinal adverse reactions | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks
  Evaluate using the "Metformin Adverse Reaction Assessment Form"，The scale consists of six items related to dyspepsia symptoms. Each item has a minimum score of 0, indicating no symptoms, and a maximum score of 3, representing symptoms that affect daily life. The higher the score, the more obvious the symptoms are and the worse the outcome.
Medication Adherence | 12 weeks, 24 weeks
  Medication adherence is evaluated by actual dosage, required dosage and medication treatment rate.
  Medication treatment rate: assesses the continuous treatment rate of metformin in both groups, the rate of continuous treatment at different dosages, the dropout rate.
  Continuous treatment rate: refers to the number of people who have been treated with metformin for 12 weeks or 24 weeks / total number of people.
  Continuous different dosage treatment rate: includes the continuous treatment rate of metformin at 1500mg/day and 2000mg/day doses, referring to the number of people who have been treated with metformin at 1500mg/day or 2000mg for 12 weeks or 24 weeks / total number of people.
  Discontinuation rate: refers to the number of people who discontinued metformin treatment at 12 weeks or 24 weeks during follow-up / total number of people.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No